CLINICAL TRIAL: NCT01123369
Title: Spectralis HRA+OCT Imaging of the Retina With Autofluorescence in Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Dr. Esther Bowie, Medcial University of South Carolina
Other Study IDs: SEI 10-001; HR#18890 (Other: Medical University of SC)
Record Dates: First submitted 2010-03-25; First posted 2010-05-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the retinal and choroidal thickness in patients with sickle cell disease compared to age, race matched population without sickle cell disease to allow a better understanding of the clinical manifestations of sickle cell retinopathy. The purpose of this research study is to evaluate the relationship between sickle cell disease and the eye. The research study is recruiting African American population with or without Sickle Cell Disease. The investigator in charge of this study is Dr E. Bowie. Approximately 60 subjects of both sexes will be enrolled at the Medical University of South Carolina.

DETAILED DESCRIPTION:
About 10% of African Americans have an abnormal hemoglobin gene. About 8% of African Americans are heterozygous for Hb S. In the United States, sickle cell anemia primarily occurs in the black population, with approximately 0.2% of African American children afflicted by this disease. The prevalence in adults is lower because of the decrease in life expectancy. The Storm Eye Institute at the Medical University of South Carolina (MUSC) is uniquely situated geographically and epidemiologically to study the interaction between sickle cell disease and the retina. The frequency of sickle cell trait (Hb AS) in African-Americans of Charleston County is 16%, twice the national average of 8% in African-Americans. This is thought to be due to the autosomal recessive inheritance of sickle cell disease, and the genetic roots and relative isolation of the Sea Island Gullah population (Pollitzer 1999).

Variations in the alteration of the amino acid sequence on the globin chain produce variations in the disease's expression. The four forms of the disease are often referred to by their genotype: sickle cell trait (AS), sickle cell anemia (SS), sickle cell disease (SC) and sickle cell thalassemia (SThal).

Systemically, the sickle cell anemia variation (SS) produces the most symptoms. With respect to the eye, the sickle cell disease mutation (SC) produces the most effects.

The widely accepted pathogenesis for sickle cell retinopathy is vasoocclusion that leads to retinal hypoxia, ischemia, infarction, neovascularization, and fibrovascularization. In sickle cell anemia, the amino acid substitution valine for glutamate occurs on the beta chain at the sixth position. This substitution, combined with conditions that may promote sickling (ie, acidosis, hypoxia), triggers the deoxygenated Hb S to polymerize, making the erythrocyte rigid. This rigidity is partially responsible for the vasoocclusion.

Vasoocclusion also is in part due to the interaction between sickled cells and the vascular endothelium. The adherence of sickled cells to the endothelium triggers an inflammatory process with the release of inflammatory agents. The result of this cascade is vascular stasis, hemolysis, and vasoocclusion of the capillary beds.

Classically, posterior segment changes are classified by either nonproliferative sickle retinopathy (NPSR) or proliferative sickle retinopathy (PSR). In NPSR, the retinal changes do not involve neovascularization as they do in PSR. The use of Spectralis HRA+OCT gives us visualization of the individual layers of the retina to determine if there are underlying changes not seen clinically in the gross ophthalmic posterior segment exam. This knowledge will aid the care of African-Americans with sickle cell disease to enable greater understanding of the ocular disease progression leading to earlier eye screenings, possible novel treatments and ultimately visual loss prevention.

ELIGIBILITY:
Inclusion Criteria:

* SUBJECTS approximately 60 subjects of both sexes of African American race with or without sickle cell disease.

Patient Inclusion Criteria:

* Subjects MUST fulfill the following conditions to qualify for enrollment into the trial
* Twelve years of age or older.
* Patients diagnosed with sickle cell disease (n=40) and an age, race matched control group of subjects (n=20) without sickle cell disease. Sickle disease is defined as a genetic blood disease due to the presence of an abnormal form of hemoglobin, namely hemoglobin S. It includes four genotypes: sickle cell trait (AS), sickle cell anemia (SS), sickle cell disease (SC) and sickle cell thalassemia (SThal). Patients with any of these genotypes will be included.
* Willing and able to comply with scheduled visit and other study procedure

Exclusion Criteria:

* Subject must not have a history of prior intraocular retinal surgery, prior laser photocoagulation, cryotherapy, active ophthalmic disease or abnormality (e.g. blepharitis, corneal infection), clinical evidence of trauma (including scarring).
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Pregnant and nursing mothers.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 60 subjects of both sexes of African American race with or without sickle cell disease.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Patient Care | 6 months
  The use of Spectralis HRA+OCT gives us visualization of the individual layers of the retina to determine if there are underlying changes not seen clinically in the gross ophthalmic posterior segment exam. This knowledge will aid the care of African-Americans with sickle cell disease to enable greater understanding of the ocular disease progression leading to earlier eye screenings, possible novel treatments and ultimately visual loss prevention

CONTACTS AND LOCATIONS:
Overall Officials: Esther M Bowie, MD, Principal Investigator — Medical University of South Carolina, Storm Eye Institute
Locations (2):
- United States (2):
  - Medical University of South Carolina, Storm Eye Institute, Charleston, South Carolina
  - MUSC Storm Eye Institute, Charleston, South Carolina